CLINICAL TRIAL: NCT04655352
Title: Single Center, Clinical Trial Examining the Safety and Tolerability of a Bacillus Subtilis Probiotic in Healthy Adult Volunteers in a Single-Blind Design
Brief Title: Safety and Tolerability of Bacillus Subtilis MB40 in Healthy Adult Volunteers
Status: Completed | Type: Observational
Sponsor: BIO-CAT Microbials, LLC (Industry)
Collaborators: Prism Research LLC (Unknown)
Responsible Party: Sponsor
Organization: BIO-CAT, Inc. (Industry)
Other Study IDs: BCT-100-000
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Healthy Participants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bacillus subtilis MB40: 1-week placebo (maltodextrin and excipients) lead-in followed by MB40 intervention
  Interventions: Dietary Supplement: Bacillus subtilis MB40

INTERVENTIONS:
Dietary Supplement: Bacillus subtilis MB40 — 1-week placebo (maltodextrin and excipients) lead-in followed by 250 mg capsule (5 billion CFU/capsule) administered twice daily for 21 days
  Other Names: OPTI-BIOME MB40

SUMMARY:
This study is a single-blind, placebo-lead in design examining the safety and tolerability of a probiotic, Bacillus subtilis MB40. Subjects received a 7-day placebo BID lead-in and a 21-day BID course of Bacillus subtilis MB40. GI questionnaires and Bristol stool charts along with evaluation of any medically significant changes, based on physical examination findings, clinical laboratory tests and vital signs assessments were used to determine the safety and tolerability of MB40.

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy adult volunteers aged 18 to 55 years.
2. BMI of 18 to 32 kg/m2 (inclusive)
3. Have no clinically significant findings on screening evaluations (clinical, laboratory)
4. If female, participant is not of child bearing potential, which is defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR

   Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:
   * Hormonal contraceptives (stable for 1 month) including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner (shown successful as per appropriate follow-up)
5. Able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

1. History or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, or psychiatric disorders.
2. Current or recent history (<30 days prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection.
3. Frequent GERD, indigestion, nausea, or vomiting (1 or more days per week).
4. Frequent abdominal pain/cramps or bloating (1 or more days per week).
5. Frequent constipation, diarrhea, or alternating constipation/diarrhea (1 or more days per week).
6. Abdominal pain before bowel movements that is relieved with defecation (most bowel movements).
7. Abdominal complaints often worsened by worry or tension (1 or more days per week).
8. Medical diagnosis of esophagitis, gastritis, ulcers, inflammatory bowel disease, gastrointestinal cancer, celiac disease, or irritable bowel syndrome.
9. Recent gastrointestinal bleeding (hematemesis, hematochezia, melena in past 3 months) or anemia in the past 3 months.
10. Unintentional weight loss of 10 lbs or more in the past 3 months.
11. Screening GI Questionnaire Score of ≥ 4 for any single item.
12. Current clinically significant viral infection
13. History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin
14. Resting heart rate less than 45 bpm or greater than 100 bpm.
15. History of unstable ischemic heart disease or uncontrolled hypertension (blood pressure >150/90 mm Hg)
16. History of stomach or intestinal surgery, except that appendectomy and/or cholecystectomy will be allowed.
17. Presence of a malabsorption syndrome possibly affecting drug/Product absorption (e.g., Crohn's disease or chronic pancreatitis)
18. History of alcoholism or drug addiction within 1 year prior to Screening, or current alcohol or drug use that, in the opinion of the investigator, will interfere with the subject's ability to comply with the dosing schedule and study evaluations.
19. Use of any tobacco-containing or nicotine-containing products (including cigarette, pipe, cigar, chewing tobacco, nicotine patch, or nicotine gum) more frequently than 50 cigarettes per week within 2 months prior to Screening or > 20 per week from screen through the end of the study
20. Current treatment or treatment within 30 days or 5 half-lives (t ½) prior to the first dose of study product with another investigational product or current enrollment in another investigational drug protocol at the time of screening.
21. Use of any over-the-counter, prescription, non-prescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations), within 7 days prior to study entry, unless deemed acceptable by the Investigator.
22. Use of greater that 2 units per day of alcohol-containing or caffeine-containing foods or beverages within 72 hours prior to study entry and throughout the duration of the study.
23. Donation of blood in excess of 500 ml within 4 weeks prior to study entry or of plasma within 2 weeks prior to Screening.
24. Receipt of blood products within 3 months prior to study entry.
25. Subjects who, in the opinion of the investigator, are unable or unlikely to comply with the dosing schedule and study evaluations.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Human volunteers meeting eligibility criteria listed above.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2015-12-17 (Actual); Study Completion 2015-12-17 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | 4 weeks
  GI Questionnaire and weekly in person assessment of adverse events

SECONDARY OUTCOMES:
Weekly mean of daily frequency of GI symptoms | 4 weeks
  GI symptom frequency and severity questionnaire
Weekly mean of daily severity of GI symptoms | 4 weeks
  GI symptom frequency and severity questionnaire

OTHER OUTCOMES:
Frequency of bowel movements | 4 weeks
  Bristol Stool Chart questionnaire
Incidence of clinically significant abnormal vital signs | Screening and day 29
Incidence of clinically significant abnormal complete blood panel | Screening and day 29

CONTACTS AND LOCATIONS:
Overall Officials: Mark Matson, MD, Study Director — Prism Research LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spears JL, Kramer R, Nikiforov AI, Rihner MO, Lambert EA. Safety Assessment of Bacillus subtilis MB40 for Use in Foods and Dietary Supplements. Nutrients. 2021 Feb 25;13(3):733. doi: 10.3390/nu13030733. PMID 33668992